CLINICAL TRIAL: NCT02668601
Title: Maternal Gestational Diabetes in Hispanic Youth: Obesity and Insulin Resistance
Brief Title: Maternal GDM in Hispanic Youth: Risk for Obesity
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Kathleen Page, Assistant Professor of Medicine, University of Southern California
Other Study IDs: HS-10-00465
Record Dates: First submitted 2015-05-11; First posted 2016-01-29 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Diabetes, Gestational; Obesity; Insulin Resistance; Insulin Secretion
Keywords: Gestational Diabetes Mellitus; Childhood Obesity; Offspring
MeSH Terms: conditions — Diabetes, Gestational; Obesity; Insulin Resistance; Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- GDM Exposed: Children exposed to gestational diabetes in utero
- Non-GDM Exposed: Children not exposed to gestational diabetes in utero

SUMMARY:
Our studies are aimed at examining effects of intrauterine exposure to GDM on metabolic risks in Hispanic children. Our primary hypothesis predicts that intrauterine exposure to GDM will be associated with one or more of three critical factors involved in the development of diabetes: 1) increased adiposity, 2) insulin resistance, and 3) decreased beta cell function in Hispanic children when compared to non-exposed children matched for ethnicity, age, gender, and Tanner stage. In a subset of this cohort, we will also examine the effects of intrauterine exposure to gestational diabetes on the brain pathways that regulate appetite and body weight in children ages 6 to 15 years old.

DETAILED DESCRIPTION:
Obesity rates have increased dramatically over the last two decades, particularly in children. Obesity is a major risk factor for type 2 diabetes (T2D), and there is a disproportionate prevalence of obesity and T2D in people of Hispanic origin. While a number of factors contribute to the development of obesity and T2D there is compelling evidence suggesting a profound role of the diabetic in utero environment. Epidemiological studies show that exposure to maternal diabetes in utero is associated with a significant risk of developing obesity and diabetes later in life. Provocative studies in animal models suggest that metabolic imprinting resulting from exposure to the altered metabolic milieu of diabetes in pregnancy leads to abnormalities in the development of specific fetal tissues, including the hypothalamus and pancreatic islets. Based on these findings, the goal of this research is to test the hypothesis that exposure to maternal gestational diabetes mellitus in utero results in changes during intrauterine development that mediate increased risk for obesity and diabetes. Through our ongoing studies on the genetics of type 2 diabetes we have access to hundreds of Hispanic offspring of well characterized GDM and control mothers. We are, therefore, in the unique position to perform mechanistic studies examining effects of intrauterine exposure to GDM on metabolic risks in Hispanic children and adolescents. Our primary hypothesis predicts that intrauterine exposure to GDM will be associated with one or more of three critical factors involved in the development of diabetes: 1) increased adiposity, 2) insulin resistance, and 3) decreased beta cell function in Hispanic children when compared to non-exposed children matched for ethnicity, age, gender, and Tanner stage.

To examine the effects of exposure to GDM on brain pathways involved in the regulation of energy homeostasis, we will perform additional functional magnetic resonance imaging (fMRI) studies in a subset of the larger cohort.

ELIGIBILITY:
Inclusion Criteria:

* Offspring between the ages of 4 and 18 years old who were born to women who participated in the BetaGene Study.

Exclusion Criteria:

* Offspring < 4 or > 18 years of age;
* gestation < 36 weeks at birth;
* significant medical illness and/or current use of medication known to influence glucose tolerance or BMI.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: GDM exposed and non-exposed Hispanic offspring of singleton pregnancies between the ages of 4 to 18 years old. Offspring are the children of women with a history of GDM or with normal glucose levels during pregnancy who participated in the BetaGene Study. Normal glucose levels during pregnancy are defined as 1-hour 50g glucose challenge test <120 mg/dl. GDM diagnosis is defined as two or more abnormal values on 3-h 100-g diagnostic OGTT. GDM defined by American Diabetes Association Criteria in place from 2003-2008.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2010-08; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Adiposity | Day 1
  BMI (z-score) and total body fat
insulin sensitivity | Day 2
  OGTT
insulin secretion | Day 2
  OGTT
hypothalamic CBF | Day 3
  fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Page, MD, Principal Investigator — University of Southern California